CLINICAL TRIAL: NCT03260751
Title: A 12-week, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Zingiber Officinale Roscoe Extract on Body Fat
Brief Title: Efficacy and Safety of Zingiber Officinale Roscoe Extract on Body Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WJ-BF-ZO
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zingiber officinale Roscoe extract 200 mg (Experimental): 2 cap/day, 800 mg/cap for 12 weeks
  Interventions: Dietary Supplement: Zingiber officinale Roscoe extract 200 mg
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zingiber officinale Roscoe extract 200 mg — 2 cap/day, 800 mg/cap for 12 weeks
  Arms: Zingiber officinale Roscoe extract 200 mg
Dietary Supplement: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Zingiber officinale Roscoe extract on body fat.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. Forty subjects were randomly divided into Zingiber officinale Roscoe extract 200 mg or placebo group. The investigators measured Body Fat Mass, Percent Body Fat, Fat Free Mass, weight, and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 65 years,
* BMI 25~29.9 kg/m2
* subjects giving written informed consent

Exclusion Criteria:

* Significant variation in weight(more 10%) in the past 3 months
* Cardiovascular disease, e.g. arrhythmia, heart failure, myocardial infarction, and patient with pacemaker
* History of disease that could interfere with the test products or impede their absorption, such as gastrointestinal disease or gastrointestinal surgery
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnancy or breast feeding etc,.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Changes of body fat mass | Baseline and 12 week
  Body fat mass was measured in study baseline and 12 week

SECONDARY OUTCOMES:
Changes of percent body fat | Baseline and 12 week
  Percent body fat was measured in study baseline and 12 week
Changes of fat free mass | Baseline and 12 week
  Fat Free Mass was measured in study baseline and 12 week
Changes of weight | Baseline and 12 week
  Weight was measured in study baseline and 12 week
Changes of body mass index | Baseline and 12 week
  Body mass index was measured in study baseline and 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided